CLINICAL TRIAL: NCT07392203
Title: Role of (Saline- Glycerin) Rectal Enema in Treatment of Fecal Incontinence in Children
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Souzan ALi Mohamed, Resident of pediatric surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-12-13MS
Record Dates: First submitted 2026-01-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anorectal Malformation
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective, single-arm, single-centre interventional study by rectal enema using saline and glyceri (Experimental): Prospective, single-arm, single-centre interventional study conducted in the Pediatric Surgery Department, Sohag University Hospitals. The protocol adheres to contemporary bowel-management frameworks for pediatric fecal incontinence with daily retrograde enemas and radiographic/clinical titration.
  Interventions: Procedure: Rectal enema using saline and glycerin mixture once daily

INTERVENTIONS:
Procedure: Rectal enema using saline and glycerin mixture once daily — Rectal enema using saline & glycerin for treatment of fecal incontinence in children

SUMMARY:
Using saline glycerin mixture once daily in children with fecal incontinence to reach aclean child without fecal accidents the next day.

DETAILED DESCRIPTION:
Child lies on Lt lateral position. Foley catheter inserted to thr rectum and inflated Instillation of saline glycerin mixture. Child hold it for 15 minutes Foley catheter removed Child stay in bathroom for 45 min

ELIGIBILITY:
InclusioChildren ≥3 and ≤16 years with Fecal incontinence (≥1 episode/week) due to corrected anorectal malformation (ARM), Hirschsprung disease after pull-through, perineal trauma, spinal anomalies/neurogenic bowel, or functional constipation with overflow incontinence.

Ability to participate in a structured bowel-management regimen at home.

Caregiver availability for training and daily administration. n Criteria:

- Age <3 years. symptomatic anal stricture, or other anatomic issues requiring surgical correction before bowel management.

Current enterocolitis, Active proctitis, painful fissure with bleeding, or severe perianal dermatitis precluding safe catheterization.

Chronic kidney disease, unstable cardiac disease, or known electrolyte imbalance.

Hypersensitivity/intolerance to glycerin; prior severe reaction to enemas. Stoma in situ or ACE dependence (separate pathway).

Exclusion Criteria:

-

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of clean days (no stool accidents) during days 7-14 of titration and at week 4. | Follow up after 4 weeks and after 12 weeks
Proportion of clean days (no stool accidents) during days 7-14 of titration and at week 4. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided